CLINICAL TRIAL: NCT02714270
Title: A Randomized Clinical Trial of Paperless Versus Modified World Health Organization Partograph in Management of First Stage of Labour
Brief Title: Paperless Partograph for Management of Low Risk Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WHOP-PP
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Normal Labor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified partograph (Active Comparator): routine modified partograph
  Interventions: Procedure: modified partograph
- paperless partograph (Active Comparator): paperless partograph with no graph paper
  Interventions: Procedure: paperless partograph

INTERVENTIONS:
Procedure: modified partograph
  Arms: modified partograph
Procedure: paperless partograph
  Arms: paperless partograph

SUMMARY:
Paperless partograph is a technique used for monitoring the progress of labor before delivery, and arriving at the accurate time to intervene for ensuring a safe delivery.

The study will be carried out to find out the effectiveness of paperless partograph in management of labor and its effect on maternal and neonatal outcomes

ELIGIBILITY:
Inclusion criteria:

1. Age: 18 to 40 years
2. Gestational age 38-42 weeks
3. Singleton pregnancy
4. Vertex presentation
5. Women who will accept to participate in the study

Exclusion criteria:

1. Malpresentation
2. Induced labour
3. Multiple pregnancy
4. Medical diseases with pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 370 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Duration of active phase of labor | 12 hours
  calculated in hours between cervical dilatation more than 3 cm till fully dilated

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes